CLINICAL TRIAL: NCT02196168
Title: A Randomized Phase II Trial of Cisplatin With or Without Wee1 Kinase Inhibitor AZD1775 (MK-1775) for First-line Treatment of Recurrent or Metastatic Squamous Cell Cancer of the Head and Neck (RM-SCCHN)
Brief Title: Cisplatin With or Without WEE1 Inhibitor MK-1775 in Treating Patients With Recurrent or Metastatic Head and Neck Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inadequate accrual rate
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NCI-2014-00759; NCI-2014-00759 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHL-088; NCI 9416; PHL-088 (Other: University Health Network Princess Margaret Cancer Center P2C); 9416 (Other: CTEP); N01CM00032 (NIH); NCT01935037 (obsolete NCT alias)
Record Dates: First submitted 2014-07-18; First posted 2014-07-21 (Estimated); Results first posted 2017-05-03 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-03

CONDITIONS: Recurrent Hypopharyngeal Squamous Cell Carcinoma; Recurrent Laryngeal Squamous Cell Carcinoma; Recurrent Laryngeal Verrucous Carcinoma; Recurrent Lip and Oral Cavity Squamous Cell Carcinoma; Recurrent Metastatic Squamous Cell Carcinoma in the Neck With Occult Primary; Recurrent Nasal Cavity and Paranasal Sinus Squamous Cell Carcinoma; Recurrent Oral Cavity Verrucous Carcinoma; Recurrent Oropharyngeal Squamous Cell Carcinoma; Squamous Cell Carcinoma Metastatic in the Neck With Occult Primary; Stage IV Hypopharyngeal Squamous Cell Carcinoma; Stage IVA Laryngeal Squamous Cell Carcinoma; Stage IVA Laryngeal Verrucous Carcinoma; Stage IVA Lip and Oral Cavity Squamous Cell Carcinoma; Stage IVA Nasal Cavity and Paranasal Sinus Squamous Cell Carcinoma; Stage IVA Oral Cavity Verrucous Carcinoma; Stage IVA Oropharyngeal Squamous Cell Carcinoma; Stage IVB Laryngeal Squamous Cell Carcinoma; Stage IVB Laryngeal Verrucous Carcinoma; Stage IVB Lip and Oral Cavity Squamous Cell Carcinoma; Stage IVB Nasal Cavity and Paranasal Sinus Squamous Cell Carcinoma; Stage IVB Oral Cavity Verrucous Carcinoma; Stage IVB Oropharyngeal Squamous Cell Carcinoma; Stage IVC Laryngeal Squamous Cell Carcinoma; Stage IVC Laryngeal Verrucous Carcinoma; Stage IVC Lip and Oral Cavity Squamous Cell Carcinoma; Stage IVC Nasal Cavity and Paranasal Sinus Squamous Cell Carcinoma; Stage IVC Oral Cavity Verrucous Carcinoma; Stage IVC Oropharyngeal Squamous Cell Carcinoma; Tongue Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Lymphoid Interstitial Pneumonia; Tongue Neoplasms | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; adavosertib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (WEE1 inhibitor MK-1775, cisplatin) (Experimental): Patients receive WEE1 inhibitor MK-1775 PO BID for 5 doses beginning on day 1 and cisplatin IV over 1 hour on day 1.
  Interventions: Drug: Cisplatin; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: WEE1 Inhibitor AZD1775
- Arm II (placebo, cisplatin) (Active Comparator): Patients receive placebo PO BID for 5 doses beginning on day 1 and cisplatin IV over 2 hour on day 1.
  Interventions: Drug: Cisplatin; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Placebo

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (placebo, cisplatin)
Drug: WEE1 Inhibitor AZD1775 — Given PO
  Other Names: AZD-1775; AZD1775; MK-1775; MK1775
  Arms: Arm I (WEE1 inhibitor MK-1775, cisplatin)

SUMMARY:
This randomized phase II trial studies how well cisplatin with or without WEE1 inhibitor MK-1775 works in treating patients with head and neck cancer that has come back or has spread to other parts of the body. Drugs used in chemotherapy, such as cisplatin, may prevent tumor cells from multiplying by damaging their deoxyribonucleic acid (DNA), which in turn stops the tumor from growing. WEE1 inhibitor MK-1775 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether cisplatin is more effective with or without WEE1 inhibitor MK-1775 in treating patients with head and neck cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the overall response rate assess the efficacy of MK-1775 (WEE1 inhibitor MK-1775) in combination with cisplatin to cisplatin alone in patients with recurrent or metastatic squamous cell carcinoma of the head and neck (SCCHN) as per overall response rate (using Response Evaluation Criteria in Solid Tumors [RECIST] criteria version [v]1.1).

SECONDARY OBJECTIVES:

I. Assess secondary measures of efficacy (progression free survival at 6 months and 12 months, overall survival rate at 12 months).

II. Assess measures of efficacy by tumor protein (p)53 status. III. Evaluate safety and tolerability. IV. Explore predictive and pharmacodynamic biomarkers.

OUTLINE:

SAFETY RUN-IN: Patients receive WEE1 inhibitor MK-1775 orally (PO) twice daily (BID) for 5 doses beginning on day 1 and cisplatin intravenously (IV) over 1 hour on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive WEE1 inhibitor MK-1775 PO BID for 5 doses beginning on day 1 and cisplatin IV over 1 hour on day 1.

ARM II: Patients receive placebo PO BID for 5 doses beginning on day 1 and cisplatin IV over 2 hour on day 1.

In both arms, courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed SCCHN that is recurrent and/or metastatic and not amendable to curative therapy by surgery or radiation; SCCHN originating from the following sites are eligible: oral cavity, oropharynx, larynx, hypopharynx and paranasal sinus; for patients with a diagnosis of SCCHN of unknown origin, their eligibility must be reviewed and approved by the principal investigator
* No prior systemic chemotherapy or WEE1 kinase inhibitor therapy for metastatic or recurrent disease will be allowed; patients are permitted to have received prior systemic chemotherapy as a part of the initial multimodality treatment for locally advanced disease if this treatment was completed more than 6 months prior to enrollment
* Patients must have disease amenable to biopsy and must be medically fit to undergo a biopsy
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 10 mm with computed tomography (CT) scan; indicator lesions must not have been previously treated with surgery, radiation therapy or radiofrequency ablation unless there is documented progression after therapy
* Patients must have completed any previous surgery or radiotherapy >= 4 weeks prior to enrollment
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (Karnofsky > 60%)
* Life expectancy of greater than 12 weeks
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 × institutional upper limit of normal
* Prothrombin time (PT)/partial thromboplastin time (PTT)/international normalized ratio (INR) =< 1.5 upper limit of normal (ULN)
* Creatinine within normal institutional limits OR calculated creatinine clearance >= 60 mL/min/1.73 m^2 for patients with levels above institutional normal using modified Cockcroft-Gault
* Cardiac function: 12-lead electrocardiogram (ECG) with normal tracing, or non-clinically significant changes that do not require medical intervention; corrected QT (QTc) interval is to be < 470 msec
* Women of childbearing potential and men must be surgically sterilized, practicing abstinence, or agree to use 2 birth control methods prior to study entry and for the duration of study participation including up to 30 days after the last dose of MK-1775; the 2 methods of birth control can be either 2 barrier methods or a barrier method plus a hormonal method to prevent pregnancy; the following are considered adequate barrier methods of contraception: diaphragm or sponge, and condom; other methods of contraception such as copper intrauterine device or spermicide may be used; appropriate hormonal contraceptives will include any registered and marketed contraceptive agent that contains an estrogen and/or a progestational agent (including oral, subcutaneous, intrauterine, or intramuscular agents); should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Past or current malignancy other than SCCHN, except for:

  * Cervical carcinoma stage 1B or less
  * Non-invasive basal cell and squamous cell skin carcinoma
  * Malignant melanoma with a complete response of a duration of > 10 years
  * Radically treated prostate cancer (prostatectomy or radiotherapy) with normal prostate specific antigen (PSA), and not requiring ongoing anti-androgen hormonal therapy
  * Other cancer diagnosis with a complete response of duration of > 5 years
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MK-1775 or cisplatin
* Patients who are unable to take oral medications and/or who have a clinical or radiological diagnosis of bowel obstruction are ineligible
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, active peptic ulcer disease, myocardial infarction within 6 months prior to entry, congestive heart failure, symptomatic congestive heart failure, active cardiomyopathy, unstable angina pectoris, cardiac arrhythmia, uncontrolled hypertension or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with MK-1775
* Human immunodeficiency virus (HIV)-positive patients are ineligible
* Patients taking the following prescription or non-prescription drugs or other products (i.e. grapefruit juice) are ineligible: sensitive cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) substrates, CYP3A4 substrates with a narrow therapeutic index, moderate to potent inhibitors/inducers of CYP3A4; patients would be eligible if the medications can be discontinued two weeks prior to day 1 of dosing and withheld throughout the study until 2 weeks after the last dose of study medication

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Winquist, Principal Investigator — University Health Network Princess Margaret Cancer Center P2C
Locations (3):
- Canada (3):
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (WEE1 Inhibitor MK-1775, Cisplatin) | Arm II (Placebo, Cisplatin)
Started | 6 | 0
Completed | 6 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (WEE1 Inhibitor MK-1775, Cisplatin) | Arm II (Placebo, Cisplatin) | Total
Number analyzed (Participants) | 6 | 0 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 3 |  | 3
  >=65 years | 3 |  | 3
Age, Continuous [Median (Full Range); unit: years] | 66 [56 to 84] |  | 66 [56 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 5 |  | 5
Region of Enrollment [Number; unit: participants]
  Canada | 6 |  | 6

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (Complete Plus Partial Response) Using RECIST Criteria v1.1
Description: Per Response Evaluation Criteria in solid Tumors (RECIST1.1) Target lesions are assessed as Complete Response(CR), Disappearance of all target lesions; Partial Response (PR),30% decrease in the sum of the diameters of target lesions; Progressive Disease (PD), At least a 20% increase (minimum 5 mm) from smallest sum (nadir); Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. Nontarget lesions are assessed as Complete Response (CR), Disappearance of all non-target lesions; Non-CR/Non-PD, Persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits; Progressive Disease (PD),Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions; Overall Response(OR); PR=CR+non-CR/non-PD,SD=SD+non-PD; PD=PD+presence of any non-target lesions
Time Frame: Up to 1 year
Measure: Number; unit: Participants
Arm/Group | Arm I (WEE1 Inhibitor MK-1775, Cisplatin) | Arm II (Placebo, Cisplatin)
Number analyzed (Participants) | 6 | 0
Participants | 0 |

2. Secondary Outcome: Incidence of Adverse Events Using the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: Gr 3, Gr 4 and Gr 5 AEs at least possibly related to study drug
Time Frame: Up to 1 year
Measure: Number; unit: adverse events
Arm/Group | Arm I (WEE1 Inhibitor MK-1775, Cisplatin) | Arm II (Placebo, Cisplatin)
Number analyzed (Participants) | 6 | 0
adverse events | 13 |

3. Secondary Outcome: Levels of Pharmacodynamic Biomarkers
Description: Predictors of clinical outcomes will be investigated using logistic regression, Cox proportional hazards regression and/or generalized estimating equations as appropriate. Descriptive statistics and plotting of data will be used to better understand potential relationships.
Time Frame: Pre-dose, at 4-8 hours on day 3 or 20-24 hours on day 4
Population: No data are available as decision was made by PI not to do the analysis due to small number of patients
Arm/Group | Arm I (WEE1 Inhibitor MK-1775, Cisplatin) | Arm II (Placebo, Cisplatin)
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

4. Secondary Outcome: Levels of Predictive Biomarkers
Description: as for outcome 3
Time Frame: Up to day 4 of course 1
Population: No data are available as decision was made by PI not to do the analysis due to small number of patients.
Arm/Group | Arm I (WEE1 Inhibitor MK-1775, Cisplatin) | Arm II (Placebo, Cisplatin)
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

5. Secondary Outcome: Overall Survival
Description: Estimated in each group by the Kaplan Meier method and differences between groups will be calculated by the log rank test. Hazard ratios for each group will be estimated using the Cox Regression model.
Time Frame: 12 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (WEE1 Inhibitor MK-1775, Cisplatin) | Arm II (Placebo, Cisplatin)
Number analyzed (Participants) | 6 | 0
months | 0.21 [0.01 to 0.60] |

6. Secondary Outcome: Progression Free Survival
Description: Progression-free survival (PFS) is defined as the duration of time from start of treatment to time of progression (20% increase in the sum of the longest diameter of target lesions or a measurable increase in a non-target lesion, or the appearance of new lesions) or death, whichever occurs first.
Time Frame: Time from start of treatment to time of progression or death, whichever occurs first, assessed at 6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (WEE1 Inhibitor MK-1775, Cisplatin) | Arm II (Placebo, Cisplatin)
Number analyzed (Participants) | 6 | 0
months | 2.88 [0.99 to NA] — The upper limit for Measure of Dispersion was 'not reached' for this study |

7. Secondary Outcome: Progression Free Survival
Description: as for outcome 5
Time Frame: Time from start of treatment to time of progression or death, whichever occurs first, assessed at 12 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (WEE1 Inhibitor MK-1775, Cisplatin) | Arm II (Placebo, Cisplatin)
Number analyzed (Participants) | 6 | 0
months | 2.88 [0.99 to NA] — The upper limit for Measure of Dispersion was 'not reached' for this study |

ADVERSE EVENTS:
Arm/Group | Arm I (WEE1 Inhibitor MK-1775, Cisplatin) | Arm II (Placebo, Cisplatin)
Serious Adverse Events (participants affected / at risk) | 4/6 | 0/0
Other Adverse Events (participants affected / at risk) | 6/6 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (WEE1 Inhibitor MK-1775, Cisplatin) (N=6) | Arm II (Placebo, Cisplatin) (N=0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0 (0)
lymphocyte count decreased (Investigations) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 3 | 0
white blood cell decreased (Investigations) | 2 | 0
neutrophil count decreased (Investigations) | 2 | 0
Generalized Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (WEE1 Inhibitor MK-1775, Cisplatin) (N=6) | Arm II (Placebo, Cisplatin) (N=0)
Anemia (Blood and lymphatic system disorders) | 4 | 0
Lymphocyte count decreased (Investigations) | 2 | 0
Neutrophil count decreased (Investigations) | 2 | 0
white blood cell decreased (Investigations) | 2 | 0
hypophosphatemia (Investigations) | 2 | 0
alkalosis (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Generalized Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less